CLINICAL TRIAL: NCT01143610
Title: A New Regenerative Therapeutic Approach for Root Coverage: a Randomized Clinical Trial
Brief Title: A New Therapeutic Approach for Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Adriana Campos Passanezi SantAna, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 115-2007
Record Dates: First submitted 2010-04-30; First posted 2010-06-14 (Estimated); Results first posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-06

CONDITIONS: Gingival Recession
Keywords: Root coverage; Graft; Soft tissue; Periodontal regeneration
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Newly forming bone (Experimental): Miller class I or II deep recessions treated by the newly forming bone technique.
  Interventions: Procedure: Newly forming bone technique for root coverage
- Subepithelial connective tissue graft (Active Comparator): Miller class I or II deep recessions treated by subepithelial connective tissue graft.
  Interventions: Other: Subepithelial connective tissue graft for root coverage.

INTERVENTIONS:
Procedure: Newly forming bone technique for root coverage — A granulation tissue will be obtained 21-25 days after the creation of an alveolar socket and grafted to receptor site.
  Other Names: Bone granulation; NFBG
  Arms: Newly forming bone
Other: Subepithelial connective tissue graft for root coverage. — A subepithelial connective tissue graft will be used for the treatment of Miller class I or II deep recessions.
  Other Names: SCTG
  Arms: Subepithelial connective tissue graft

SUMMARY:
Different surgical techniques have been proposed for root coverage, showing varying results especially in areas of deep recessions. The aim of this study is to evaluate the effectiveness of the newly forming bone technique (NFB)as an alternative treatment for Miller class I or II deep recessions, requiring regeneration of lost periodontal tissues. Sample should be comprised of patients aged 18-45 years, both genders, presenting at least one site with marginal tissue recession >4mm. Patients will be randomly assigned to either one of the groups, based on treatment technique: newly forming bone (NFB) or subepithelial connective tissue graft (SCTG). Clinical examinations will be performed by a single blinded examiner at baseline, 1, 3, 6 and 9 months after surgery. Intra-group analysis will be performed by one way analysis of variance for repeated measures. Inter-group analysis will be performed by unpaired t-test for each of evaluation periods.

DETAILED DESCRIPTION:
Both gender patients presenting Miller class I or II recession defects >4mm were selected. Patients were randomly assigned to treatment groups: newly forming bone graft (NFBG) or subepithelial connective tissue graft (SCT). Patients were treated in the period of February 2008 and March 2008 and monitored during 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with at least one tooth presenting marginal tissue recession equal to or greater than 4mm in depth and one edentulous area or tooth to be extracted.

Exclusion Criteria:

* Smokers
* Pregnants
* Use of anti-convulsants, anti-hypertensives, cyclosporine or hormones
* Use of antibiotics for the last 6 months
* Patients under treatment for medical conditions or presenting systemic disorders that would impair treatment results (e.g.: uncontrolled diabetes mellitus)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana P Sant'Ana, DDS PhD, Principal Investigator — School of Dentistry at Bauru, University of São Paulo; Bruna R Ferraz, DDS, Principal Investigator — School of Dentistry at Bauru, University of São Paulo
Locations (1):
- School of Dentistry at Bauru-USP, Discipline of Periodontics, Bauru, São Paulo, Brazil

REFERENCES:
- See also: School of Dentistry at Bauru, University of São Paulo site information — http://www.fob.usp.br

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients both genders, 18-45 years, showing at least one site with gingival recession should attend the Graduation Clinics of Periodontics, School of Dentistry at Bauru-USP, from October to December 2007 for enrollment in a new treatment protocol.
Pre-assignment Details: Participants were excluded from the study prior to group assignement in cases of pregnancy, diagnosis of systemic disease or if the patient quit participating.
Period: Overall Study
Arm/Group | Newly Forming Bone | Subepithelial Connective Tissue Graft
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Newly Forming Bone | Subepithelial Connective Tissue Graft | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41 (4.24) | 41.5 (2.67) | 41.26 (3.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  Brazil | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Root Coverage
Description: Percentage of root coverage determined by: [area covered]/[total area to be covered] x 100 (in %)
Time Frame: Baseline, 9 months post-operatively
Population: The unity of analysis was the site, since each participant contributed with more than one site for treatment
Measure: Mean (Full Range); unit: percentage of area covered
Units Other Than Participants: sites
Arm/Group | Newly Forming Bone | Subepithelial Connective Tissue Graft
Number analyzed (Participants) | 7 | 8
Number analyzed (sites) | 35 | 30
percentage of area covered | 66 [40 to 90] | 73 [50 to 100]

2. Secondary Outcome: Gain of Clinical Attachment Level
Description: Investigation of clinical attachment level, probing depth and reduction of recession depth
Time Frame: 9 months post-operatively
Population: The unit of analysis was the site, since each participant contributed with more than one site to be treated
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: sites
Arm/Group | Newly Forming Bone | Subepithelial Connective Tissue Graft
Number analyzed (Participants) | 7 | 8
Number analyzed (sites) | 35 | 30
mm | 3.74 (0.26) | 2.95 (0.19)

ADVERSE EVENTS:
Arm/Group | Newly Forming Bone | Subepithelial Connective Tissue Graft
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No